CLINICAL TRIAL: NCT06210581
Title: Comparison of the Effects of Internet-Based and Supervised Exercise Programs in People With Multiple Sclerosis
Brief Title: The Effects of Internet-Based and Supervised Exercise Programs in People With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tahire Basak Demir, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC2023-04
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: Balance; Multiple Sclerosis; Exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): The treatment sessions will be terminated by performing relaxation exercises combined with stretching and breathing exercises.
  Interventions: Other: Supervised Exercise Program Group
- Group II (Other): Patients who are in the internet-based exercise program group will register cite ''https://www.telenororehab.com /'' which is web- based physiotherapy program for exercises.
  Interventions: Other: Internet Based Exercise Program Group

INTERVENTIONS:
Other: Supervised Exercise Program Group — The exercise programs will performed with the physiotherapist. The treatment programs of the patients will start with warm-up exercises and continue with aerobic exercises. Strengthening exercises will be performed in lying, sitting and standing positions. Body weight or free weight will be used for strengthening exercises. Balance exercises will be performed in sitting and standing positions and will be performed with or without support according to the patients conditions. The treatment sessions will be terminated by performing relaxation exercises combined with stretching and breathing exercises.
  Arms: Group I
Other: Internet Based Exercise Program Group — Patients who are in the internet-based exercise program group will register cite ''https://www.telenororehab.com /'' which is web- based physiotherapy program for exercises. After the first evaluation patients will be given a username and password to log in to the system.
  Before starting the exercise programs, the pages on how patients can log in to the system, how they can reach the physiotherapist through the system and how they can find individual exercise programs will be shown before the study. After logging in to their own pages, patients will be able to access video-based exercise programs that have been specially prepared for them. Patients in the Internet-based exercise program group will also be given the same exercise programs as the supervised exercise program group. The entry-exit times of patients to the system and the duration of maintaining exercise programs will be controlled from the administrator section on the system.
  Arms: Group II

SUMMARY:
The main aim of this study is resarch and compare the effects of supervised exercise programs and internet-based exercise programs, which have started to benefit from their effects in recent years, known for not requiring conditions such as transportation distance, cost and time, on motor disorders and quality of life in people with multiple sclerosis (MS). This study conducting for develop a new perspective on conventional physiotherapy and rehabilitation practices. Our study will be performed in people with MS with a high EDSS score, is seen as an important contribution for the literature.

DETAILED DESCRIPTION:
The groups were included in exercise programs of 16 sessions in total, twice a week for 8 weeks. Exercise programs will consist of warm-up, aerobic exercises, strengthening exercises, balance exercises, breathing exercises, cooling and relaxation exercises. Exercise programs will be created by the physiotherapist and arranged every 2 weeks according to the patients' conditions. Patients who do not participate in the program 2 times in a row will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MS by a neurologist
* Being between ages of 18-65
* Not having had an attack in the last 3 months
* The score of Expanded Disability Status Scale (EDSS) is 5.5- 7.5
* Not participating in a another physiotherapy and rehabilitation program
* Having internet access

Exclusion Criteria:

* Pregnancy
* Severe cognitive impairment that effects participating to rehabilitation
* The cardiopulmonary disease that will prevent aerobic exercise
* Having a major hearing and/or vision problem
* Having a major speech disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-05-29 (Estimated); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
2 Minutes Walk Test (2MWT) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  This test is performed for the assessment of walking endurance. The patient is informed about the test before starting the test. The distance that a person walks along a 25-meter corridor in 2 minutes is calculated in meters. During the test, patients who have tiredness and shortness of breath can have a rest.

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a scale used for the evaluation of fatigue in MS patients. It consists of a total of 9 questions. A minimum of 1 and a maximum of 7 points can be scored from each question. The minimum score that can be obtained from the test is 9 the maximum score is 63. High scores mean that fatigue has increased. Validity and reliability studies have been conducted in Turkish MS patients of the FSS.
12 Item MS Walking Scale (MSWS- 12) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is used for evaluating walking ability in MS patients. This scale evaluates the limitations faced by MS patients in walking in the last two weeks. Situations such as loss of balance during walking, running, going up and down stairs, standing and walking, slowing down of walking are questioned. It is a Likert-type scale consisting of 12 questions. Each question score to between 1 and 5 points. The high scores indicate that the ability to walk is affected or that there is difficulty in walking.
Modified Falls Efficacy Scale (MFES) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  The MFES aims to assess the impact of a person's fear of falling on daily living activities. MFES is consist of 14 items (10 indoor and 4 outdoor activitiy) and every question can score to 0-10. Low scores indicates high fear of falling.
Canadian Occupational Performance Measure (COPM) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  COPM evaluates the activities that a person has difficulty doing in daily life between 1-10 points as activity performance and satisfaction score. At least one, up to 5 activities can be written, resulting in a total performance and satisfaction score. These scores are divided by the number of activities written, resulting in an average performance and satisfaction score. A validity and reliability study of the scale was conducted in individuals with MS.
Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  ): It is a scale that assess the quality of life in MS patients. MusiQoL has 9 subgroups and 31 questions. During the evaluation, patients are asked to take into account their condition for the last 4 weeks. The answers to each question and the points that can be obtained; It is never/ Never (0 points), Rarely/ A little (1 point), Sometimes/ A little (2 points), Often/ A lot (3 points), Always/ Too much (4 points). The lowest score that can be taken from the scale is 0, the highest score is 124, and a high score indicates a low quality of life.
The Multiple Sclerosis Impact Scale (MSIS- 29) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  ): It is a scale consisting of a total of 29 items that evaluate the consequences of symptoms and limitations caused by MS. It is a Likert type scale consisting of 5 points that evaluates the severity of symptoms such as fatigue, tremor, muscle spasm, personal care activities, sleep problems, concentration disorders. 1= having no problems at all, 2= having very few problems, 3= having moderate problems, 4= having severe problems, 5= having very severe problems. A total of at least 29 and a maximum of 145 points. A high score indicates a high amount of yeti loss.
Berg Balance Scale (BBS) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  BBS developed for the functional assessment of balance in adults. it consists of 14 divisions. Each section is scored 0 to 4 points. 0= cannot do the task, 4= does it independently. A minimum of 0 and a maximum of 56 points can be scored. Low scores indicate a balance disorder. 0-20 points indicate a balance disorder, 21-40 points indicate an acceptable balance, 41-56 points indicate the presence of a good balance. There is a validity and reliability study of the scale in MS patients.
5 Times Sit to Stand Test (5TSTS) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  The patient is asked to sit on a chair with his arms crossed in a way to hold the other shoulders. The patient is told to sit down and get up 5 times as fast as possible. The test is terminated as soon as the person's pelvic area comes into contact with the chair. Increased time indicates a disturbed balance. The test has validity in MS patients.
Timed 25- Foot Walk (T25- FW) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is used for the evaluation of walking speed in MS patients. the patient is asked to walk the distance of 7.62 meters (25 steps) as fast as possible. The time is calculated in seconds. The timed 25-step walking test is known as a very suitable test for evaluating walking speed in MS patients.
Timed Get up and Go Test (TUG) (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  TUG used to measure the balance and functional capacities of MS patients. The patient is asked to sit on a chair and a distance of 3 meters is determined. It is requested that the patient be with a shoe that he always uses. The patient is asked to get up from the chair, walk this distance and sit in the chair again. At this time, the time is kept in seconds by the stopwatch. High test times means reduce balance and high risk of falling. Its use in individuals with MS has been shown to be reliable and valid.

CONTACTS AND LOCATIONS:
Overall Officials: Yonca ZENGINLER YAZGAN, Study Chair — Istanbul University-Cerrahpasa Faculty of Health Science; Murat KURTUNCU, Study Chair — Istanbul University Faculty of Medicine Department of Neurology
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patient's information will not be shared.

REFERENCES:
- See also: Article — http://doi.org/10.7224/1537-2073.2015-006
- See also: Article — http://doi.org/10.4274/jmsr.galenos.2021.2021-10-3
- See also: Article — http://doi.org/10.7224/1537-2073.2017-046
- See also: Article — http://doi.org/10.23736/S1973-9087.18.05366-2
- See also: Article — http://doi.org/10.1055/S-0038-1649502